CLINICAL TRIAL: NCT03146481
Title: Effect of Pre-operative Aceclofenac on the Anesthetic Efficacy of Inferior Alveolar Nerve Block in Patients With Symptomatic Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: Pre-operative Aceclofenac on the Anesthetic Efficacy of IANB in Symptomatic Irreversible Pulpitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nermeen AwadAllah Abbas Ibrahim, Principal Investigator, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CEBD-CU-2015-5-145
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Irreversible Pulpitis
Keywords: Anesthetic efficacy, Irriversible pulpitis, Aceclofenac
MeSH Terms: interventions — aceclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aceclofenac (Experimental): Aceclofenac 100 mg tablet
  Interventions: Drug: Aceclofenac
- placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aceclofenac — Aceclofenac 100 mg tablet given one hour before starting the root canal treatment
  Other Names: Bristaflam
  Arms: Aceclofenac
Other: Placebo — Placebo tablet given one hour before starting the root canal treatment
  Arms: placebo

SUMMARY:
The aim of this randomized, double-blinded, controlled study is to evaluate the effect of pre-operative oral aceclofenac on the success of the inferior alveolar nerve block with 2% Mepivacaine containing 100,000 Epinephrine for patients with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
* The aim of this randomized, double-blinded, controlled study is to evaluate the effect of pre-operative oral aceclofenac on the success of the inferior alveolar nerve block with 2% Mepivacaine containing 100,000 Epinephrine for patients with symptomatic irreversible pulpitis.
* Patients will be clinically and radiographically examined and their eligibility will be assessed and preoperative pain will be measured using Heft-Parker VAS. Eligible patients will be treated in one visit.
* Patients will be randomly assigned to one of 2 groups: experimental group (taking a 100 mg of Aceclofenac) and the control group (taking a placebo tablet). Each tablet will be taken one hour before starting treatment. After 15 minutes of the initial inferior alveolar nerve block (IANB), the teeth will be examined using a cold pulp sensitivity test; in case of no or mild pain, the treatment will be initiated otherwise, additional IANB will be administered.
* During root canal treatment, no to mild pain response will be considered success. In case of failure, supplemental anesthesia will be administrated.

ELIGIBILITY:
Inclusion Criteria:

* Patients in good health (American Society of Anesthesiologists Class I or Class II).
* Patients having symptomatic irreversible pulpitis in one of their mandibular molars
* Age is 18 years or older.
* Patients who can understand Heft- Parker Visual Analogue Scales.
* Patients able to sign informed consent.

Exclusion Criteria:

* Patients allergic to aceclofenac or Mepivacaine.
* Pregnant or nursing women.
* Patients having active pain in more than one molar in the same quadrant.
* Administration of analgesics within 12 h before the administration of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Anesthetic success | intraoperative
  Success of mandibular inferior alveolar nerve block anesthesia during access cavity preparation and instrumentation which will be measured with Heft-parker VAS in which no or mild pain will be considered as anesthetic success and moderate or severe pain will be considered as anesthetic failure.

SECONDARY OUTCOMES:
Pain on injection of inial IANB | intraoperative
  Pain on injection of inial IANB will be measured with Heft-Parker VAS

CONTACTS AND LOCATIONS:
Overall Officials: Nermeen A Abbas, Postgraduate, Principal Investigator — Cairo University; Suzan AW Amin, PhD, Study Director — Cairo University; Shaimaa Gawdat, PhD, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramachandran A, Khan SI, Mohanavelu D, Kumar KS. The efficacy of pre-operative oral medication of paracetamol, ibuprofen, and aceclofenac on the success of maxillary infiltration anesthesia in patients with irreversible pulpitis: A double-blind, randomized controlled clinical trial. J Conserv Dent. 2012 Oct;15(4):310-4. doi: 10.4103/0972-0707.101881. PMID 23112474
- [Background] Jena A, Shashirekha G. Effect of preoperative medications on the efficacy of inferior alveolar nerve block in patients with irreversible pulpitis: A placebo-controlled clinical study. J Conserv Dent. 2013 Mar;16(2):171-4. doi: 10.4103/0972-0707.108209. PMID 23716973